CLINICAL TRIAL: NCT01547572
Title: Psychological Preparation for Colorectal Surgery: Impact of Video Education. A Randomised Trial
Brief Title: Psychological Preparation for Colorectal Surgery: Impact of Video Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ihedioha, Ugo, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: IhediohaU
Record Dates: First submitted 2012-02-27; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Use of Video Education; Colorectal Surgery
Keywords: Video education; Enhanced recovery; Reducing hospital stay; Improving patient satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group (Experimental): The study group will get a video and leaflet on enhanced recovery.
  Interventions: Procedure: The study group will get a video and leaflet on enhanced recovery
- Control group (No Intervention): The control group will receive a leaflet only.
  Interventions: Procedure: The control group will receive a leaflet only

INTERVENTIONS:
Procedure: The study group will get a video and leaflet on enhanced recovery — The study group will get a video and leaflet
  Arms: Study group
Procedure: The control group will receive a leaflet only — The control group will receive a leaflet only
  Arms: Control group

SUMMARY:
Since the introduction and favourable early results of enhanced recovery programmes more than a decade ago, such programmes have become increasingly popular following major surgery. Many elements of these programmes are based on solid evidence and derived from published trials. These programmes optimize different factors to reduce the stress of surgery with the aim of improving patient outcome and speed up recovery after surgery. Key factors prior to surgery are conditioning of expectations and optimizing associated disease. Strategies during the operation include use of short-acting anaesthetic (sleeping) agents, maintenance of normal temperatures and minimal access surgery (keyhole surgery).

Care after surgery is optimized with appropriate analgesia (pain killers), early mobilisation (walking) and early feeding. This combined approach reduces hospital stay to 2-4 days. There is also evidence that the improvements resulting from the implementation of an enhanced recovery programme do not cause significant deterioration in quality of life or transfer costs to another component of health care.

The relative contribution of each of the single elements in the enhanced recovery programme remains uncertain. Good patient information gives confidence and improves overall outcome. No studies have examined the impact of video education on recovery.

The aim of this study is to explore the use of video information provision for patients participating in an enhanced recovery programme.

DETAILED DESCRIPTION:
TRIAL DESIGN:

A randomised controlled trial of the impact of video education in preparing patients for surgery within an enhanced recovery programme. Patients will be recruited from Leicester General Hospital and will include everyone undergoing colorectal(bowel) surgery. A standard protocol (treatment regime) is in place for all such patients. The primary end-point (main aim) will be length of hospital stay. Secondary end-points (other factors to be considered) will be patient satisfaction scores (using SF-36 outcomes in patients) and will allow the investigation of the potential implications of incorporating video education of enhanced recovery programmes into routine clinical practice.

METHODS:

All surgeons treating the patients in this trial will have a specialist interest in colorectal (bowel) surgery. All patients undergoing planned bowel surgery for benign (non-cancerous) and malignant (cancerous) disease will be eligible. Patients who cannot speak or understand english will have interpreters. Ethics approval will be sought and informed (signed) consent both for the surgery and the trial will be obtained. The study group will get a video and leaflet and the control group will receive a leaflet only. Randomisation (Division into groups) will be done using a table of random numbers to assign each study participant to a group. The consultants and registrars in charge of taking care of patients after their surgery will not be aware of which group patients belong to and a standard discharge criteria will be used (Patients for discharge should have normal observations and normal bloods results, free from lines in the hands and tubes in the waterworks, be fully mobile (walking), able to get in and out of bed unaided and dress independently. Hospital stay will be recorded in days from the time the patient is admitted to hospital. Social reasons for non-discharge such as delay in setting up home help etc will be recorded for both groups of patients.

The time to passage of flatus (wind from the back passage) and bowel motion (stool) will be recorded for each patient. Episodes of nausea and vomiting (sickness) will also be recorded as will any complication up to 30 days after surgery.

All patients will complete a questionnaire (SF-36) prior to surgery and at 3 months after surgery to assess satisfaction and return to normal activities such as leisure activities and work in the home etc.

DETAILS OF THE ENHANCED RECOVERY PROGRAMME:

Preoperative preparation (Prior to surgery) All patients will be allowed free fluids (liquids) and high calorie (energy) drinks for up to 2 hours before operation. Patients undergoing right hemicolectomy (right sided bowel surgery) will not receive bowel preparation (bowel cleansing) while those having left sided surgery will receive phosphate enema on the morning of surgery. All patients will receive antibiotic and DVT (blood clot) prophylaxis.

All patients will have baseline blood tests.

Anaesthesia (During surgery)

A standardised anaesthetic (sleeping) protocol (treatment regime) will be used for all patients. Normal temperature will be maintained throughout surgery and all operations will be carried out through the smallest incision (cut) necessary to complete the procedure. No nasogastric tubes (stomach tubes) will be used.

Postoperative pain and analgesia (Pain relief after surgery) Analgesia(Pain relief) will be provided in both groups for 48 hours via PCA (patient controlled pain relief), epidural (pain relief via injection at the back) or TAPP block (pain relief via injection on the belly).

Paracetamol will be administered concurrently with NSAIDS (non steroidal drugs) and tramadol for breakthrough pain once morphine is discontinued. Visual analogue (facial expression) pain scores at rest and movement will be measured daily until discharge. All analgesia (pain relieving drugs) used after surgery will be recorded including any discharge medication.

Diet and Fluids:

Oral fluids will be pushed immediately postoperatively (after surgery) in both groups. In addition, protein drinks and normal food will be encouraged in both groups from day 1. All lines in the arm will be removed by day 2 unless there is a clinical reason to maintain them. Both groups will have daily blood tests.

All patients will have chest physiotherapy (exercises) and will be encouraged to mobilise (walk) on day one with the help of a nurse or physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing planned bowel surgery for benign (non-cancerous) and malignant (cancerous) disease will be eligible

Exclusion Criteria:

* Patients who are unfit for surgery or undergoing emergency surgery will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The primary end-point ( main aim ) will be length of hospital stay. | Participants will be assessed for the duration of their hospital stay which is an average of 7 days.
  Hospital stay will be recorded in days from the time the patient is admitted to
  hospital.

SECONDARY OUTCOMES:
Secondary end-points will be patient satisfaction scores | Measured 3 months after discharge
  Secondary end-points ( other factors to be considered ) will
  be patient satisfaction scores ( using SF-36 outcomes in patients )

CONTACTS AND LOCATIONS:
Locations (1):
- Leicester General Hospital, Leicester, Leicestershire, United Kingdom